CLINICAL TRIAL: NCT03130283
Title: Study Design of the Empirical Evaluation of the AISBE Program in Catalonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carme Hernandez, Senior Research IDIBAPS, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SELFIE-HH/ED
Record Dates: First submitted 2017-04-10; First posted 2017-04-26 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Unrecognized Condition
Keywords: Acute patients; Exacerbated chronic patients

STUDY DESIGN:
Intervention Model Description: quasi experimental study design with propensity score matching
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Hospitalization (Active Comparator): Visit every day at home
  Interventions: Other: Home Hospitalization
- Conventional Hospitalization (Placebo Comparator): Review Clinical History
  Interventions: Other: Conventional Hospitalization

INTERVENTIONS:
Other: Home Hospitalization — Visit every 24 hours
  Arms: Home Hospitalization
Other: Conventional Hospitalization — No intervention
  Arms: Conventional Hospitalization

SUMMARY:
The project has a threefold aim: (i) Assessment of Home Hospitalization and Early Discharge (HH/ED) deployment at Hospital Clinic over a period of 10 years (2006-2015) as a preliminary analysis fo the second aim (ii) Large scale deployment of HH/ED and Transitional Care services; and, (iii) Population-based study on cost-effectiveness of integrated care services in the urban healthcare sector of Barcelona-Esquerra (540.000 inhabitants). The central hypothesis is that the approach will show safety and effectiveness with high level of user's acceptance and health value generation leading to sustainability of the service.The preliminary data indicate that HH/ED shows potential to strengthen care coordination between highly specialized hospital-based care and home-based services involving different levels of complexity. The need for appropriately designed transitional care services has been identified as the best option, not only for an efficient transference of patients from hospital to the community after hospital discharge, but as a way to overcome well identified limitations for generalization of community-based integrated care services.

AISBE is a population-based health initiative aiming at deployment of integrated care in one urban healthcare sector (Barcelona-Esquerra, 540.000 inhabitants) in the city of Barcelona. Within this initiative, the HH/ED program carried out by Hospital Clinic provides home-based hospitalization. Moreover, the program aims to implement transitional care strategies for optimal discharge.

The current document describes three studies: (Study 1) Analysis of the period 2006-2015; (Study 2) Program-based analysis of Home Hospitalization/Early Discharge (HH/ED) , and, (Study 3) Population-based analysis of cost-effectiveness of AISBE-based services. Study 2 is a program-based analysis of Home Hospitalization/Early Discharge (HH/ED). A quasi-experimental design. That is, a non-randomized intervention group (integrated care) will be compared with a control group (usual care) using propensity score matching wherein age, gender and health risk scoring will be main matching variables. The population-based evaluation will be done using registry data obtained from the Catalan Health Surveillance System (CHSS).

The protocol evaluation follows a Triple Aim approach considering pre-defined outcome variables for: a) health and well-being, b) experience with care, and c) costs.

DETAILED DESCRIPTION:
AIMS: 1) To evaluate the HH/ED as mainstream service during the last decade (2006-2015); 2) To assess healthcare value generation of during the process of large scale deployment of the HH/ED program including generation of information useful for further refinement of transitional care in AISBE; and, 3) To assess the cost-effectiveness of AISBE's integrated care services using a population-based approach. These studies will contribute to refine three core aspects of the ongoing services; that is, a) Service evaluation; b) Health risk assessment and service selection; and, c) Service workflow definition and execution.

Study 1 - It evaluates both characteristics and outcomes of the process of HH/ED deployment from 2006 to 2015 without a control group.

Study 2 - Since late 2016, HH/ED is offered as a first choice for hospitalization to patients admitted in the Emergency room of Hospital Clinic. The current program has potential for 36 home-based admissions on a 24x7 day basis. The study will cover all patients admitted in the program (estimated 1,500 candidates) using both registry data and electronic medical records. Moreover, a subset of 200 consecutive HH candidates admitted through the Emergency room at Hospital Clinic will be selected using a 1:4 ratio. They will perform a complete study adding administration of standardized questionnaires carried out during HH/ED admission, one-month and three month after HH/ED discharge.

The intervention group will receive the standard HH/ED service and it will be compared with a control group that will include the same number of patients (n=200) under conventional hospitalization. The control group will be selected from those patients admitted in the Emergency room of the Hospital Clinic, but transferred to Hospital Sagrat Cor (within AISBE) for conventional hospitalization. Inclusion of the control group will also follow 1:4 ratio. Matching between intervention and control groups will be periodically assessed by groups of 10 patients.

The study design, as described, does not include Early Discharge patients included from highly specialized programs carried out at Hospital Clinic. Consequently, an additional HH/ED group of 100 patients from those programs will be also characterized (without control group) in order to properly identify the needs of this subset of patients for transitional care.

Finally, the population-based study (Study 3) will assess the Barcelona-Esquerra as intervention group will be compared with data from the other three healthcare sectors from the city of Barcelona, taken as control groups, because they do no have well identified integrated care programs.

ELIGIBILITY:
Inclusion Criteria:

* Living in his/her house within the healthcare sector
* Having caregiver during 24h per day
* Having phone at home
* Signing written acceptance to participate in the study

Exclusion Criteria:

* High risk of severe clinical deterioration not treatable at home, as assessed by best medical judgment
* Admission in a short stay unit; and, iii) severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Costs | 30 days
  Health Care Cost

SECONDARY OUTCOMES:
Health and well-being | 30 days
  Hospital admissions
Experience with care | 30 days
  Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Carme Hernandez, PhD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic. Integrated Care Unit, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez C, Herranz C, Baltaxe E, Seijas N, Gonzalez-Colom R, Asenjo M, Coloma E, Fernandez J, Vela E, Carot-Sans G, Cano I, Roca J, Nicolas D. The value of admission avoidance: cost-consequence analysis of one-year activity in a consolidated service. Cost Eff Resour Alloc. 2024 Apr 15;22(1):30. doi: 10.1186/s12962-024-00536-1. PMID 38622593
- [Derived] Herranz C, Gonzalez-Colom R, Baltaxe E, Seijas N, Asenjo M, Hoedemakers M, Nicolas D, Coloma E, Fernandez J, Vela E, Cano I, Molken MR, Roca J, Hernandez C. Prospective cohort study for assessment of integrated care with a triple aim approach: hospital at home as use case. BMC Health Serv Res. 2022 Sep 7;22(1):1133. doi: 10.1186/s12913-022-08496-z. PMID 36071439
- See also: NEXTCARE is an innovation project belonging to the Healthcare Ris3Cat community lead by Biocat which officially starts on October 2016 — http://www.nextcarecat.cat
- See also: SELFIE (Sustainable intEgrated care modeLs for multi-morbidity: delivery, FInancing and performancE) is a Horizon2020 EU project — http://www.selfie2020.eu/